CLINICAL TRIAL: NCT07143409
Title: Fungal Vascular Graft Infections, French Multicenter Retrospective Study
Acronym: FUNGIVAS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/025
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Fungal Infection; Vascular Grafting
Keywords: vascular graft infection; vascular endograft infection; fungi; Candida
MeSH Terms: conditions — Mycoses; Torulopsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: epidemiology and medical treatment strategies — Analysis of the epidemiology and medical and surgical treatment strategies for fungal IPEV in France between January 2013 and January 2023

SUMMARY:
Fungal vascular graft and endograft infections (VGEIs) are rare but life-threatening infections. Best therapeutic management is unknown. This study retrospectively gathers fungal VGEIs from 12 university hospital centers in France over a 10 year's period in order to describe their epidemiology, clinical features, therapeutic management and outcomes. Focusing on Candida spp. VGEIs, we aim to determine prognosis factors associated with therapeutic management

DETAILED DESCRIPTION:
Fungal vascular graft and endograft infections (VGEIs) are rare but life-threatening infections. Candida spp. is the most frequent fungal agent. Main risk factor is prostheto-digestive fistula. Best therapeutic management is unknown. The aim of FUNGIVAS study is to describe epidemiology, clinical features, therapeutic management and outcomes of fungal VGEIs and determine prognosis factors associated with therapeutic management. This study retrospectively gathers fungal VGEIs from 12 university hospital centers in France from January 2013 to January 2023. Patients will be identified from mycology laboratories that have diagnosed the fungal infection on a vascular sample. Demographic, clinical, biological, imaging and outcome data will be collected using a secure and anonymous questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old with diagnosis of vascular graft and endograft infections (VGEI) in accordance to MAGIC criteria with diagnosis of proven invasive fungal infection according to EORTC criteria.
* No opposition to re-use data.

Exclusion Criteria:

* Patient previously treated for fungal VGEI
* Patient with suspected VGEI diagnosis based solely on prosthesis implantation in an infected site
* Poor understanding of French.
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fungal infection on a vascular sample
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality | Year 1
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Rate of mortality | Month 1
  Rate of all-cause mortality
Fungal vascular graft and endograft infections-related mortality | Month 1, Year 1
  Fungal vascular graft and endograft infections-related mortality
Rate of cure | Year 1
  Rate of cure, defined as : alive and without therapeutic failure (non-control of infection requiring repeat surgery or modification of anti-infective treatment)
Rate of sequelae | Year 1
  Rate of sequelae

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No